CLINICAL TRIAL: NCT04423822
Title: Contributions and Limitations of the Stress Test on the Prediction of Cardiovascular Events in a High-risk Firefighter Population
Brief Title: Stress Test on the Prediction of Cardiovascular Events in a High-risk Firefighter Population
Acronym: FIRE-PREV
Status: Terminated | Type: Observational
Why Stopped: failure to recruit
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Other Study IDs: 19CH235; 2020-A00270-39 (Other: ANSM)
Record Dates: First submitted 2020-06-08; First posted 2020-06-09 (Actual); Last update posted 2022-01-11 (Actual); Status verified 2021-12

CONDITIONS: High Cardiovascular Risk; Firefighter
Keywords: firefighter; high cardiovascular risk; stress tests
MeSH Terms: interventions — Exercise Test

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Firefighter: Firefighter with high cardiovascular risk
  Interventions: Other: stress test

INTERVENTIONS:
Other: stress test — endurance capacity

SUMMARY:
If the risk of myocardial infarction in activity is widely demonstrated to date for firefighters, and the realization of a stress test in those at high cardiovascular risk included in the practice habits, no study has evaluated the contributions and limits of the realization of a stress test in this specific population of firefighters at high cardiovascular risk for the prediction of cardiovascular events.

DETAILED DESCRIPTION:
The professional practice of firefighting presents risks specific, especially cardiovascular. In the United States 30% of Firefighter deaths are the result of a myocardial infarction that occurred while on duty. Certain occupational tasks expose firefighters to a higher risk of myocardial infarction (high physical load, inhalation of products). There is no recommendation on how to assess cardiovascular risk in French firefighters. In the absence of consensus, the Loire Departmental Fire and Rescue Service has constructed a scale for collecting cardiovascular risk factors (expert working group) to identify firefighters at high cardiovascular risk. A maintenance visit (mandatory every two years until the age of 38 and then once a year) is the best way to assess this cardiovascular risk, with a biological assessment and an electrocardiogram after the age of 40. If cardiovascular risk factors are present and the cardiovascular risk is high, the resting electrocardiogram should be supplemented by an exercise test. An exercise test can directly or indirectly quantify the endurance capacities of firefighters and reveal cardiac abnormalities sometimes absent at rest. Half of all myocardial infarctions occur without any prior symptomatology and remain totally asymptomatic, discovered during routine examinations. If the risk of myocardial infarction in activity is widely demonstrated to date for firefighters, and the realization of a stress test in those at high cardiovascular risk included in the practice habits, no study has evaluated the contributions and limits of the realization of a stress test in this specific population of firefighters at high cardiovascular risk for the prediction of cardiovascular events.

ELIGIBILITY:
Inclusion Criteria:

* Any professional or volunteer firefighter with a high cardiovascular risk attached to the Departmental Fire and Rescue Service of the Loire who has carried out an effort test between 2006 and 2014.
* Subject who received informed oral information about the study by telephone and agreed to participate in the study

Exclusion Criteria:

* Subject unable to understand the study
* Subject matter subject to a legal protection measure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: firefighters with high cardiovascular risk
Sampling Method: Probability Sample
Enrollment: 94 (Actual)
Dates: Start 2021-01-12 (Actual); Primary Completion 2021-09-18 (Actual); Study Completion 2021-09-18 (Actual)

PRIMARY OUTCOMES:
Cardiovascular morbidity | Between 2006 and 2014
  determined by occurrence of: Cardiovascular death; Myocardial infarction; stroke; Arteriopathy; Atrial fibrillation
Cardiovascular mortality | Between 2006 and 2014
  determined by occurrence of: Cardiovascular death; Myocardial infarction; stroke; Arteriopathy; Atrial fibrillation

CONTACTS AND LOCATIONS:
Overall Officials: David HUPIN, MD, Principal Investigator — CHU SAINT-ETIENNE
Locations (1):
- Centre Hospitalier Universitaire, Saint-Etienne, France

IPD SHARING:
Plan to Share IPD: No